CLINICAL TRIAL: NCT02246972
Title: BRAVEMIND: Advancing the Virtual Iraq/Afghanistan PTSD Exposure Therapy System for MST
Brief Title: BraveMind: Advancing the Virtual Iraq/Afghanistan PTSD Exposure Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Telemedicine & Advanced Technology Research Center (Other); University of Southern California (Other)
Responsible Party: Principal Investigator, Barbara O. Rothbaum, PhD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00072196
Record Dates: First submitted 2014-09-19; First posted 2014-09-23 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Trauma; Post-Traumatic Stress Disorder
Keywords: PTSD; Military sexual trauma; Veterans; Women in the military; Sexual assault
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic; Military Sexual Trauma | interventions — Virtual Reality Exposure Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VRET Immediate treatment (Experimental): Participants will be randomized to receive Virtual Reality Exposure Therapy (VRET) immediately
  Interventions: Behavioral: Virtual Reality Exposure Therapy (VRET)
- Waitlist (Active Comparator): 6 weeks standard of care, then Virtual Reality Exposure Therapy (VRET) treatment.
  Interventions: Behavioral: Virtual Reality Exposure Therapy (VRET)

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy (VRET) — 6 to 12 90-minute individual treatment sessions. During VRET sessions patients will wear a head-mounted display with stereo earphones that will provide visual and audio cues consistent with Iraqi or Afghan military scenarios or other base-related scenarios as appropriate for the individual patient.
  Other Names: VRET

SUMMARY:
The proposed study is designed to test the clinical efficacy of the BRAVEMIND military sexual trauma (MST) system in an initial feasibility and wait list clinical trial of 45 users.

The following hypotheses will be tested:

1. Virtual Reality Exposure Therapy (VRET) will be safely deliverable to persons with posttraumatic stress disorder (PTSD) due to MST as evidenced by treatment dropout rates that are similar to existing Prolonged Exposure (PE) therapy delivered in military samples (20-40%) and by the absence of any critical incidents.
2. Participants in the VRET group will show statistically and clinically meaningful reductions in PTSD and depression (PTSD Checklist-Military (PCL-M), Clinician Administered PTSD Scale (CAPS), and Patient Health Questionnaire (PHQ-9) scores and psychophysiological measures) following treatment.
3. Participants in the VRET group will show statistically and clinically meaningful reductions in PTSD and depression (PCL-M, CAPS, PHQ-9 scores and psychophysiological measures) compared to wait-list results.

DETAILED DESCRIPTION:
Pre-Treatment Assessment:

Potential subjects will be asked to provide a copy of their DD214 to verify their military service record. Once a potential participant has met all screening inclusion and exclusion criteria and consented to participate, the CAPS will be administered to determine current PTSD status.

Randomization:

Following pre-treatment assessment, patients will be randomized to receive VRET (Virtual Reality Exposure Therapy) immediately or wait 6 weeks during which time they will continue to receive usual care. Wait-listed participants will be reassessed prior to beginning their course of treatment with the Clinician Administered PTSD Scale (CAPS), PTSD Checklist-Military (PCL-M), Beck Depression Inventory-II (BDI-II), and psychophysiological measures. This pre-treatment assessment visit will last about 2-3 hours.

Therapy:

Participants will be treated once or twice per week for 6-12 sessions. VRET treatment will be limited to a minimum of 6 sessions and a maximum of 12 sessions, based upon reaching criterion of 70% symptom improvement as indicated on the PCL-M from baseline or an agreement between clinician and participant that maximum treatment response has been achieved. All sessions will be individual and weekly or twice weekly. The first session will last approximately 90 minutes and will be spent in information gathering, treatment planning, and explaining the treatment rationale to the patient. Information gathering will review the history of PTSD and their military service and will include a brief psychosocial history, including review of prior treatment.

Session 2 will discuss in vivo exposure and construct the hierarchy for in vivo exposure. The VRET sessions will last 90 minutes each. During VRET sessions patients will wear a head-mounted display with stereo earphones that will provide visual and audio cues consistent with Iraqi or Afghan military scenarios or other base-related scenarios as appropriate for the individual patient. The therapist will make appropriate comments and encourage continued exposure to the identified index trauma until anxiety has habituated. During exposure, information will be gathered on the participant's anxiety level through the use of a 0-100 Subjective Units of Discomfort (SUDs) scale. All therapists will have been trained in Prolonged Imaginal Exposure therapy (PE) followed by training in VRET by Drs. Rothbaum and Gerardi. Drs. Rothbaum and Gerardi will supervise all therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 45 males and females between ages of 18 and 65
* Participants must meet DSM-V criteria for PTSD due to military sexual trauma (MST)
* Patients must be literate in English
* Patients must be medically stable
* Participants must comprehend his or her role in the study and the risks involved

Exclusion Criteria:

* Patients with a history of mania, schizophrenia, or other psychoses
* Patients with active suicidal risk
* Patients with current alcohol or drug dependence
* Patients unable to wear the VR head mounted display
* Patients on psychotropic medications must have been on a stable dose for at least 2 months prior to beginning the study and must agree not to change their current medication regimen throughout the course of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Safely deliverable | 2 years
  Treatment dropout rates that are similar to existing PE delivered in military samples (20-40%) and by the absence of any critical incidents.
Reduction in PTSD and depression | 3 months
  Participants in the VRET group will show statistically and clinically meaningful reductions in PTSD and depression (PCL-M, CAPS, PHQ-9 scores and psychophysiological measures) following treatment.
Reduction in PTSD and depression: wait-list comparator | 6 months
  Participants in the VRET group will show statistically and clinically meaningful reductions in PTSD and depression (PCL-M, CAPS, PHG-9 scores and psychophysiological measures) compared to wait-list results.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O Rothbaum, PhD/ABPP, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States